CLINICAL TRIAL: NCT06624982
Title: Determinants of Bone Dimensional Changes After Extraction and Alveolar Ridge Preservation
Status: Recruiting | Type: Observational
Sponsor: Marquette University (Other)
Responsible Party: Principal Investigator, Vrisiis Kofina, Director, Advanced Education in Periodontics Program, Assistant Professor of Periodontics, Marquette University
Other Study IDs: HR-4787
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Alveolar Bone Grafting; Bone Healing; Tooth Extraction Site Healing; Wound Healing
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Non-molar sites with immediate post-extraction ridge expansion: Non-molar sites with an increase of buccolingual bone width immediately after tooth extraction compared to pre-extraction.
  Interventions: Other: observational study
- Non-molar sites with no immediate post-extraction ridge width change: Non-molar sites without a change in buccolingual bone width immediately after tooth extraction compared to pre-extraction.
  Interventions: Other: observational study
- Molar sites with immediate post-extraction ridge expansion: Molar sites with an increase of buccolingual bone width immediately after tooth extraction compared to pre-extraction.
  Interventions: Other: observational study
- Molar sites with no immediate post-extraction ridge width change: Molar sites without a change in buccolingual bone width immediately after tooth extraction compared to pre-extraction.
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — Observational study; alveolar ridge preservation

SUMMARY:
The main purpose of the study is to measure and localize immediate post extraction changes i.e. socket expansion versus no width change along the socket wall and identify whether the immediate post-extraction ridge width condition (expansion or no change) is a determinant of buccolingual ridge width and height changes 4 months following extraction and ridge preservation.

DETAILED DESCRIPTION:
The null hypothesis for this study is that there is no difference in bone ridge width and height changes 4 months following extraction and alveolar ridge preservation at sites that undergo immediate post-extraction socket expansion or no immediate post-extraction ridge width change. Patients of the Graduate Periodontics Clinic at Marquette University School of Dentistry scheduled for extraction, bone graft and resorbable membrane will be recruited for this study.

After providing informed consent and prior to local anesthesia and extraction, the following parameters will be recorded: age, gender, race, medical history, medications, tooth site, reason for extraction and tooth mobility. Gingival width will be recorded prior to local anesthesia and extraction, and at 4 months. Gingival thickness will be recorded after local anesthesia and prior to extraction, and at 4 months. Buccolingual ridge width and ridge height will be recorded immediately before, immediately after extraction, and at 4 months. Immediately after extraction, the following measurements will be recorded: buccal bone thickness, number of roots, root length and width, instruments used for extraction, need for flap elevation, duration of extraction, anesthetic amount, type and approach, and operator experience.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-75 years)
* Good general health (controlled conditions)
* Controlled periodontal disease
* Scheduled for single tooth extraction with bone graft placement and resorbable membrane
* Tooth to be extracted must have adjacent teeth
* Socket wall integrity

Exclusion Criteria:

* Smoking
* Pregnancy
* Active periodontal disease
* Systemic conditions that affect healing
* Lack of socket wall integrity (bone loss ≥50 %) prior to extraction, teeth with severe infection requiring pre-extraction antibiotic treatment to control infection), and contraindications for tooth extraction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for tooth extraction and alveolar ridge preservation (bone graft and membrane) in the Graduate Periodontics Clinic at Marquette University School of Dentistry.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Buccolingual ridge width | (1) After local anesthesia and before extraction, (2) immediately after extraction and (3) 4 months after extraction and alveolar ridge preservation
  Buccolingual ridge width will be measured through a stent via ridge mapping calipers. The measurement locations will be at 1mm, 3mm and 5mm from the midbuccal crest. The same measurements will be recorded at all selected time points.
Ridge height | (1) After local anesthesia and before extraction, (2) immediately after extraction and (3) 4 months after extraction and alveolar ridge preservation
  Ridge height will be measured through a stent via a periodontal probe as the distance between bone and predetermined landmarks on the stent. The measurement locations will be mesial buccal, midbuccal, distal buccal, mesial lingual, midlingual and distal lingual. The same measurements will be recorded at all selected time points.

CONTACTS AND LOCATIONS:
Overall Officials: Vrisiis Kofina, DDS, MS, Principal Investigator — Marquette University
Locations (1):
- Marquette University School of Dentistry Graduate Periodontics Clinic, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No